CLINICAL TRIAL: NCT00392535
Title: Conventional or Hypofractionated High Dose Intensity Modulated Radiotherapy for Prostate Cancer: CHHIP
Brief Title: Intensity-Modulated Radiation Therapy in Treating Patients With Localized Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000510112; ICR-CTSU-CHHIP-2006-10007; ISRCTN97182923; EU-20646
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (Active Comparator): conventional radiotherapy (74 Gy delivered in 37 fractions over 7·4 weeks)
  Interventions: Radiation: conventional radiotherapy 74 Gy delivered in 37 fractions
- Hypofractionated arm 1 (Experimental): Hypofractionated radiotherapy (60 Gy in 20 fractions over 4 weeks)
  Interventions: Radiation: hypofractionated radiation therapy 60 Gy in 20 fractions
- Hypofractionated arm 2 (Experimental): Hypofractionated radiotherapy (57 Gy in 19 fractions over 3·8 weeks)
  Interventions: Radiation: hypofractionated radiation therapy 57 Gy in 19 fractions

INTERVENTIONS:
Radiation: conventional radiotherapy 74 Gy delivered in 37 fractions
  Arms: Control arm
Radiation: hypofractionated radiation therapy 60 Gy in 20 fractions
  Arms: Hypofractionated arm 1
Radiation: hypofractionated radiation therapy 57 Gy in 19 fractions
  Arms: Hypofractionated arm 2

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. It is not yet known which schedule of intensity-modulated radiation therapy is more effective in treating patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying the side effects of three schedules of intensity-modulated radiation therapy and compares how well they work in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of conventional vs hypofractionated high-dose intensity-modulated radiotherapy in patients with localized prostate cancer.
* Determine the side effects of these regimens in these patients.
* Determine whether hypofractionated radiotherapy schedules will improve the therapeutic ratio by either improving tumor control or reducing normal tissue side effects.
* Compare acute and late treatment-related gastrointestinal and urological toxicity in these patients.
* Determine different prostate-specific antigen-related endpoints for local failure and distant metastases.
* Extend the database of patients treated to escalated doses with dose-volume histograms (DVHs) of normal tissues at risk and relate these to common toxicity endpoints.
* Develop a model to estimate normal tissue complication probability (NTCP) of rectum and bladder for hypofractionated as well as conventional dose-escalated radiotherapy schedules.

OUTLINE: This is a multicenter, randomized, pilot study. Patients are stratified according to risk of seminal vesicle involvement (low-risk vs moderate-risk or high-risk).

* Hormone therapy: Patients receive androgen-deprivation therapy comprising an injection of luteinizing hormone-releasing hormone (LHRH) agonist once monthly for 3-6 months and oral cyproterone acetate beginning the week before the first LHRH agonist injection and continuing for at least 2 weeks after each LHRH agonist injection. Within one week after the last LHRH agonist injection, patients proceed to radiotherapy.
* Radiotherapy: Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients undergo conventional high-dose intensity-modulated radiotherapy (IMRT) in 37 fractions over 7.5 weeks.
  * Arm II: Patients undergo hypofractionated high-dose IMRT in 20 fractions over 4 weeks.
  * Arm III: Patients undergo hypofractionated high-dose IMRT in 19 fractions over 3.8 weeks.

In all arms, treatment continues in the absence of unacceptable toxicity.

Quality of life is assessed periodically during study treatment.

After completion of study treatment, patients are followed periodically for up to 15 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 2,163 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate, meeting the following criteria:

  * Clinical stage T1b-T3a, N0, M0
  * Locally confined disease
  * Previously untreated disease
* Prostate-specific antigen (PSA) ≤ 30 ng/mL
* Estimated risk of seminal vesicle involvement < 30%

  * Estimated risk of seminal vesicle involvement is defined as PSA + ([Gleason score - 6] x 10) (i.e., if Gleason score ≤ 6, then PSA must be ≤ 30 ng/mL; if Gleason score = 7, then PSA must be < 20 ng/mL; if Gleason score = 8, then PSA must be < 10 ng/mL; if Gleason score = 9 or 10 patient is ineligible)

PATIENT CHARACTERISTICS:

* WHO performance status 0 or 1
* Life expectancy > 10 years (5 years for patients with poorly differentiated cancers)
* WBC > 4,000/mm^3
* Hemoglobin > 11g/dL
* Platelet count > 100,000/mm^3
* No other active malignancy within the past 5 years except basal cell carcinoma
* No hip prosthesis or fixation that would interfere with standard radiation beam configuration
* No comorbid conditions likely to impact on the advisability of radical radiotherapy (e.g., previous inflammatory bowel disease, previous colorectal surgery, significant bladder instability, or urinary incontinence)

PRIOR CONCURRENT THERAPY:

* No prior pelvic radiotherapy
* No prior radical prostatectomy
* No prior androgen-deprivation therapy
* No concurrent full anticoagulation therapy with warfarin or heparin

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3216 (Actual)
Dates: Start 2002-10-18 (Actual); Primary Completion 2015-09-08 (Actual); Study Completion 2021-06-17 (Estimated)

PRIMARY OUTCOMES:
Time to biochemical or clinical failure | Defined as the time from randomisation to biochemical failure or prostate cancer recurrence up to 5 years
  Phoenix consensus guidelines as a PSA concentration greater than nadir plus 2 ng/mL.

SECONDARY OUTCOMES:
Disease-free survival | time from randomisation to any prostate cancer-related event or death from any cause up to 15 years
Overall survival | Time from randomisation to death from any cause up to 15 years
Development of metastases | Time from randomisation to development of metastases up to 15 years
Recommencement of hormonal treatment for disease recurrence | Time from randomisation to recommencement of hormone treatment for disease recurrence up to 15 years
Acute and late side-effects | Peak and week 18 bowel and bladder side-effects

CONTACTS AND LOCATIONS:
Overall Officials: David P. Dearnaley, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (26):
- United Kingdom (26):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Addenbrooke's Hospital, Cambridge, England
  - Countess of Chester Hospital, Chester, England
  - Walsgrave Hospital, Coventry, England
  - Eastbourne District General Hospital, Eastbourne, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Ipswich Hospital, Ipswich, England
  - Clatterbridge Centre for Oncology, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Royal Marsden - London, London, England
  - Christie Hospital, Manchester, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Whiston Hospital, Prescot, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Halton Hospital, Runcorn, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southport and Formby District General Hospital, Southport, England
  - Royal Marsden - Surrey, Sutton, England
  - Warrington Hospital NHS Trust, Warrington, England
  - Worthing Hospital, Worthing, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Result] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- See also: ISRCTN registry — https://doi.org/10.1186/ISRCTN97182923